CLINICAL TRIAL: NCT06347380
Title: Usability Study of the FemPulse System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FemPulse Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP011
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-02

CONDITIONS: Overactive Bladder
Keywords: neuromodulation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Subjects receiving FemPulse System (Experimental): Subjects will receive the Ring for the treatment of their OAB symptoms
  Interventions: Device: FemPulse System

INTERVENTIONS:
Device: FemPulse System — Subjects to receive the FemPulse System consisting of a non-implanted, vaginal electrical stimulation device (Ring) and other patient accessories.

SUMMARY:
The objective of the study is to demonstrate that the FemPulse System can be used as indicated in the Instructions for Use (IFU), as applicable.

ELIGIBILITY:
Key Inclusion Criteria:

* Females, defined as a person with a uterus and cervix, ≥21 years old, with a diagnosis of OAB and symptoms for more than 6 months, as confirmed by a physician
* Able to read, comprehend, and reliably provide informed consent and study-related information.
* Willing and able to comply with study required procedures and visits (e.g., maintaining consistent medication use, fluid intake, diary completion).
* Has adequate cognitive and manual capabilities to operate the FemPulse System and other components (e.g., mobile app) as assessed by the investigator.

Key Exclusion Criteria:

* Currently pregnant, was pregnant in the past 12 months or intending to conceive during the study period.
* Plans to begin other OAB therapies or otherwise change their existing therapy regimen during the study period.
* Not an appropriate study candidate as determined by investigator.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females, defined as a person with a uterus and cervix.
Enrollment: 5 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 28 days
  Proportion of subjects reporting satisfaction with the use of the FemPulse System

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Sponsor GmbH
Locations (2):
- United States (2):
  - Holy Cross Women's Hospital, Fort Lauderdale, Florida
  - Univ. of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No